CLINICAL TRIAL: NCT02198183
Title: The Effects of Positive-pressure Ventilation on Cerebral Oxygenation and Cardiac Output in Total Shoulder Arthroplasty.
Brief Title: Total Shoulder Arthroplasty Near-infrared Spectroscopy
Acronym: TSA NIRS
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-003
Record Dates: First submitted 2014-07-16; First posted 2014-07-23 (Estimated); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Near-infrared spectroscopy: Casmed Fore-Sight Elite and Non-invasive Cardiac Output Monitor (NICOM)
  Interventions: Device: Casmed Fore-Sight Elite; Device: Non-invasive Cardiac Output Monitor (NICOM)

INTERVENTIONS:
Device: Casmed Fore-Sight Elite
Device: Non-invasive Cardiac Output Monitor (NICOM)

SUMMARY:
The purpose of this study is to measure cerebral oxygenation and cardiac output of total shoulder replacement patients undergoing general anesthesia (GA) and positive-pressure ventilation (PPV).

We hypothesize that cerebral desaturation occurs frequently during GA with PPV, but is rare during GA and spontaneous ventilation. We also hypothesize that cardiac output usually is well maintained under GA in the sitting position when epinephrine is used, but that decreased cardiac output increases the risk of cerebral desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-99 undergoing total shoulder arthroplasty
* Planned general anesthesia + brachial plexus nerve block
* Planned arterial catheter

Exclusion Criteria:

* Patients younger than 18 years older and older than 99
* Patients not intending to receive general anesthesia and peripheral nerve block
* Indication for endotracheal tube
* BMI ≥ 30
* Ejection Fraction (if known) < 50%
* Known significant restrictive or obstructive pulmonary disease
* Patients with a history of transient ischemic attack (TIA) or stroke
* Patients with recent signs or symptoms of myocardial ischemia

  * Current stress test positive for ischemia
* Intolerance to study medications
* pre-existing contraindication to regional anesthesia

  * infection at block site
  * pre-existing neurological injury to operative limb
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total shoulder arthroplasty patients who are receiving surgery at the Hospital for Special Surgery
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Friedman DJ, Parnes NZ, Zimmer Z, Higgins LD, Warner JJ. Prevalence of cerebrovascular events during shoulder surgery and association with patient position. Orthopedics. 2009 Apr;32(4):orthosupersite.com/view.asp?rID=38058. PMID 19388618
- [Background] Yadeau JT, Casciano M, Liu SS, Edmonds CR, Gordon M, Stanton J, John R, Shaw PM, Wilfred SE, Stanton M. Stroke, regional anesthesia in the sitting position, and hypotension: a review of 4169 ambulatory surgery patients. Reg Anesth Pain Med. 2011 Sep-Oct;36(5):430-5. doi: 10.1097/AAP.0b013e318228d54e. PMID 21857267
- [Background] Yadeau JT, Liu SS, Bang H, Shaw PM, Wilfred SE, Shetty T, Gordon M. Cerebral oximetry desaturation during shoulder surgery performed in a sitting position under regional anesthesia. Can J Anaesth. 2011 Nov;58(11):986-92. doi: 10.1007/s12630-011-9574-7. Epub 2011 Aug 25. PMID 21866430
- [Background] Koh JL, Levin SD, Chehab EL, Murphy GS. Neer Award 2012: cerebral oxygenation in the beach chair position: a prospective study on the effect of general anesthesia compared with regional anesthesia and sedation. J Shoulder Elbow Surg. 2013 Oct;22(10):1325-31. doi: 10.1016/j.jse.2013.01.035. Epub 2013 Apr 6. PMID 23571083

RESULTS

PARTICIPANT FLOW:
Groups:
- Near-infrared Spectroscopy: Casmed Fore-Sight Elite and Non-invasive Cardiac Output Monitor (NICOM)
  Casmed Fore-Sight Elite
  Non-invasive Cardiac Output Monitor (NICOM)
Period: Overall Study
Arm/Group | Near-infrared Spectroscopy
Started | 34
Completed | 25
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Patients that were enrolled and not excluded due to receiving an intra-operative endotracheal tube or missing data from the monitors or instruments used.
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Cerebral Desaturation Events
Description: The number of Cerebral Desaturation Events (CDE) that occured. CDE is defined as a reduction in cerebral tissue oxygen saturation of >20% from baseline that lasts for 90 seconds or longer.
Time Frame: Day of surgery
Measure: Number; unit: Number of CDE Incidences
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
Number of CDE Incidences | 0

2. Secondary Outcome: Cardiac Output (CO)
Description: Cardiac output of patients as measured in liters per minute
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
liters per minute | 5.6 (1.2)

3. Secondary Outcome: Cardiac Index (CI)
Description: Average cardiac index for patients, a measurement of how efficient the heart is pumping. Measured in liters per minute per meters squared of heart size.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
L/min/m^2 | 3 (0.5)

4. Secondary Outcome: Stroke Volume (SV)
Description: Stroke volume, the amount of blood pumped by the left ventricle of the heart with each contraction. Measured in milliliters.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
milliliters | 74 (11)

5. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: mean arterial pressure and noninvasive blood pressure will be represented as a percentage of baseline after surgery. A lower percentage is a worse outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
percent
  GA without PPV | 76 (15)
  GA with PPV | 67 (17)

6. Secondary Outcome: End Tidal Carbon Dioxide (ETCO2)
Description: a lower score is a better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
mmHg
  GA without PPV | 44 (5)
  GA with PPV | 45 (6)

7. Secondary Outcome: Intravenous Fluid Volume
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Near-infrared Spectroscopy
Number analyzed (Participants) | 25
mL | 1408 (227)

ADVERSE EVENTS:
Arm/Group | Near-infrared Spectroscopy
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes